CLINICAL TRIAL: NCT01817348
Title: Effect of Combined Intra-articular Injection of Lidocaine Plus Physiotherapy in Treatment of Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20121001R
Record Dates: First submitted 2013-01-08; First posted 2013-03-25 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Frozen Shoulder; Adhesive Capsulitis
Keywords: Adhesive capsulitis; Frozen shoulder; Shoulder pain; Intra-articular injection; Lidocaine injection; Physiotherapy; Manipulation; Stretch exercise
MeSH Terms: conditions — Bursitis; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine group (Experimental): 1% lidocaine 5ml intra-articular injection to shoulder joint + physiotherapy three times weekly
  * Injection is performed if pain during intervention equals to or greater than 7cm in a 10-cm VAS scale.
  * Injection frequency is not greater than twice per week and total injection time is limited to 10 times in the whole course
  * In each week, patient will receive 3 times of PT with or without intra-articular lidocaine injection.
  Interventions: Procedure: Lidocaine group; Other: Physiotherapy (PT)
- PT group (Placebo Comparator): - Apply to every patient, each by the same physical therapist, 3 times weekly for 3 months or till the patients gain satisfactory results.
  Interventions: Other: Physiotherapy (PT)

INTERVENTIONS:
Procedure: Lidocaine group — * Patient position: prone position with arm under the abdomen and the elbow flexed to a right angle
  * Injection with a 25-gauge, 1.5-inch long needle fitted with 3ml syringe filled with 3ml 1% lidocaine.
  Arms: Lidocaine group
Other: Physiotherapy (PT) — - Include electric therapy, hot pack, followed by stretch exercise and joint mobilization
  Other Names: Physiotherapy

SUMMARY:
1. Therapeutic exercise, especially stretch exercise and joint mobilization, remain the mainstay of conservative treatment of frozen shoulder.

   1. Nevertheless, shoulder pain during the physiotherapy reduces the treatment effect.
   2. Manipulation or arthroscopic release under general anesthesia may avoid pain during the intervention; however, increased risk of humeral shaft fracture and failure of release of pathological tissue were reported.
2. We consider intra-articular injection is a compromized way, from a practical point of veiw, to reduce the pain during physiotherapy.
3. We hypothesize that, intra-articular injection with lidocaine before joint mobilization and stretch exercise, can make the patient pain-free during physiotherapy, and the effect of combined therapy is superior to physiotherapy alone in the treatment of frozen shoulder.

DETAILED DESCRIPTION:
A randomized controlled trial to compare the effect in treatment of frozen shoulder between combined intra-articular injection with lidocaine plus physiotherapy and physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed as unilateral frozen shoulder, with the definition as more than 50% loss of passive movement of the shoulder joint relative to the non-affected side, in one or more of the three movement direction (ie. abduction in the frontal plane, forward flexion in sagittal plane, or external rotation in 0 degree of abduction)
* Duration of complaints of more than three months
* Ability to complete questionnaires in Chinese

Exclusion Criteria:

* History of shoulder fracture, dislocation, or trauma
* History of Rheumatic arthritis, tumor, or other diseases in the shoulder joints
* Receive intra-articular corticosteroid injection or manipulation therapy in shoulder joint in recent four weeks
* Pregnancy or breast feeding
* Allergic to lidocaine

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in range of motion at 3-months intervention | baseline; 1 month; 2 months; 3 months
  * Measured with a conventional goniometer by a physiotherapist, both active and passive range of motion
  * Including shoulder flexion, abduction, internal rotation, and external rotation
  * All measurements will be rounded off to the nearest five degrees
Change from Baseline in range of motion at 3 months post-intervention | baseline; 1 and 3 months after completion
  * Measured with a conventional goniometer by a physiotherapist, both active and passive range of motion
  * Including shoulder flexion, abduction, internal rotation, and external rotation
  * All measurements will be rounded off to the nearest five degrees

SECONDARY OUTCOMES:
Visual analog scale (VAS) | baseline; 1 month; 2 months; 3 months; 1 and 3 months after completion
  * Horizontal lines of 100mm, with 0 indicating no pain on the left and 100 indicating very severe pain on the right
  * Three separate visual analog scales: shoulder pain at rest, during movement, and during the night
36-Item Short-form health survey (SF-36) | baseline; 1 month; 2 months; 3 months; 1 and 3 months after completion
  * General health status measurement
  * 8 subscales for physical functioning, social functioning, role limitations (physical problems, emotional problems), mental health, vitality, pain, and general health perception
  * Each subscale generates a score from 0 to 100, with higher score indicating better health
Shoulder Rating Questionnaire (SRQ) | baseline; 1 month; 2 months; 3 months; 1 and 3 months after completion
  * Self-administered questionnaire
  * Include global assessment, pain, daily activities, recreational and athletic activities, work, satisfaction, and areas for improvement.
  * Total score ranges from a minimum of 17 points (worst) to a maximum of 100 points (best functional status)
Shoulder Disability Questionnaire (SDQ) | baseline; 1 month; 2 months; 3 months; 1 and 3 months after completion
  * For shoulder disability measurement
  * Consists of 23 symptoms that participants respond to with either "yes" or "no" or "not applicable"
  * Score ranges from 0 to 100, is the number of positive response divided by the number of answered questions multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsu WC, Wang TL, Lin YJ, Hsieh LF, Tsai CM, Huang KH. Addition of lidocaine injection immediately before physiotherapy for frozen shoulder: a randomized controlled trial. PLoS One. 2015 Feb 25;10(2):e0118217. doi: 10.1371/journal.pone.0118217. eCollection 2015. PMID 25714415